CLINICAL TRIAL: NCT04353973
Title: A Randomized Study of an eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Predisposition in Metastatic Breast, Ovarian, Prostate and Pancreatic Cancer Patients
Brief Title: Study of an eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Predisposition in Metastatic Cancer Patients
Acronym: eReach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: AstraZeneca (Industry); Fox Chase Cancer Center (Other); Basser Center for BRCA (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC 11919; IRB#833370 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2020-04-03; First posted 2020-04-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A (Experimental): Visit 1/Pre-Test Session - Standard-of-Care Pre-Test Counseling with a genetic counselor either in-person or by remote services (Telephone or Video Conferencing).
  Visit 2/Disclosure Session - Standard-of-Care Post-Test Counseling with a genetic counselor either in-person or by remote services (Telephone or Video Conferencing).
  Interventions: Other: Standard of Care
- ARM B (Experimental): Visit 1/Pre-Test Session - Standard-of-Care Pre-Test Counseling with a genetic counselor either in-person or by remote services (Telephone or Video Conferencing).
  Visit 2/Disclosure Session - Self-directed web-based eHealth result disclosure intervention.
  Interventions: Other: Standard of Care; Other: Post-Test Intervention
- ARM C (Experimental): Visit 1/Pre-Test Session - Self-directed web-based eHealth pre-test session intervention.
  Visit 2/Disclosure Session - Standard-of-Care Post-Test Counseling with a genetic counselor either in-person or by remote services (Telephone or Video Conferencing).
  Interventions: Other: Pre-Test Intervention; Other: Standard of Care
- ARM D (Experimental): Visit 1/Pre-Test Session - Self-directed web-based eHealth pre-test session intervention.
  Visit 2/Disclosure Session - Self-directed web-based eHealth result disclosure intervention.
  Interventions: Other: Pre-Test Intervention; Other: Post-Test Intervention

INTERVENTIONS:
Other: Pre-Test Intervention — Secure and accessable by private code only, the web-based intervention will provide users with a the results of their clinical genetic testing results and a detailed summary of what those results mean. Additionally, an individualized summary will also be included.
  Arms: ARM C; ARM D
Other: Standard of Care — Standard of Care with a Genetic Counselor either In-Person or by Remote Services (Telephone or Video Conferencing)
  Arms: ARM A; ARM B; ARM C
Other: Post-Test Intervention — Secure and accessable by private code only, the web-based intervention will provide users with a the results of their clinical genetic testing results and a detailed summary of what those results mean. Additionally, an individualized summary will also be included.
  Arms: ARM B; ARM D

SUMMARY:
This study aims to determine if web-based eHealth delivery of pre-test and/or post-test counseling in cancer patients and/or those at risk for cancer can provide equal or improved cognitive and affective outcomes when compared to the standard of care delivery model.

DETAILED DESCRIPTION:
Cancer genetic testing has become a standard evidence-based practice, with established risk reduction and cancer screening guidelines for genetic carriers. With FDA approval for PARP inhibitors in patients with advanced breast, ovarian, pancreatic and prostate cancer, there is an additional therapeutic rationale for testing all breast, ovarian, pancreatic and prostate cancer patients for germline genetic mutations. Yet, access to genetic specialists is limited in many area, and the traditional model of pre- and post-test counseling with a genetic professional will not support the rising indications for cancer genetic testing. Thus, there is an urgent need to consider alternative delivery models to increase access and uptake of testing, while maintaining adequate patient outcomes.

This study aims to assess if traditional pre-test (visit 1) and post-test (visit 2: disclosure) counseling delivered by a genetic counselor can be replaced with a self-directed web-based eHealth intervention to provide critical data to inform optimal ways to deliver cancer genetic testing in patients with breast, ovarian, pancreatic and prostate cancer, while maintaining quality of care and favorable cognitive, affective and behavioral outcomes.

Specific Aim 1: To determine if web-based eHealth delivery of pre-test and/or post-test counseling can provide equal or improved cognitive and affective short-term and 6-month outcomes as compared to the two-visit standard of care delivery model with a genetic counselor. The investigator's primary outcomes will be changes in knowledge and anxiety. Secondary outcomes will include uptake of testing, depression, cancer specific distress, uncertainty and health behaviors and provider time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak and understand English
* Male or Female
* A personal history of one or more of the following:

  * metastatic breast cancer
  * advanced ovarian cancer (Stage III-IV)
  * metastatic pancreatic cancer
  * metastatic prostate cancer
* Naive to previous cancer germline genetic testing

Exclusion Criteria:

* Communication difficulties such as:

  * Uncorrected or uncompensated hearing and/or vision impairment
  * Uncorrected or uncompensated speech defects
  * Uncontrolled psychiatric/mental condition or severe physical, neurological or cognitive deficits rendering individual unable to understand study goals and tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge | Baseline - Within 7 days of Visit 2
  Knowledge Scale - Score Range = 0-16 Increased change score indicates increase in knowledge (better).
Change in Anxiety | Baseline - Within 7 days of Visit 2
  Patient-Reported Outcomes Measurement Information Systems (PROMIS) - Score Range = 4-20 Decreased score change indicates a decrease in anxiety (better).

SECONDARY OUTCOMES:
Change in Depression | Baseline - Within 7 days of Visit 2
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Score Range = 4-20 Decreased score change indicates a decrease in depression (better).
Change in Cancer Specific Distress | Baseline - Within 7 days of Visit 2
  Impact of Events Scale (IES) - Score Range = 0-40 Decreased score change indicates a decrease in distress (better).
Change in Uncertainty | Within 7 days of Visit 2 - 6-Month Follow-Up
  Multi-dimensional Impact of Cancer Risk Assessment Questionnaire (MICRA) - Score Range = 0-85 Decrease in score change indicates a decrease in uncertainty (better).
Change in Health Behaviors | Within 7 days of Visit 2 - 6-Month Follow-Up
  Change in treatment plan and communication of results - Yes/No
Provider Time | Within 7 days of Standard of Care V1
  Time (minutes) provider spends per study participant
Provider Time | Within 7 days of Standard of Care V2
  Time (minutes) provider spends per study participant
Frequency of Uptake of Testing | Within 7 days of Visit 1
  Testing uptake per arm - Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KT, McLeod B, Egleston B, Brown S, Howe S, Fetzer D, Gutstein L, Cacioppo C, Clark D, Domchek SM, Ebrahimzadeh J, Falcone D, Ofidis D, Griffin H, Mim R, Hernandez S, Fleisher L, Karpink K, Selmani E, Tahsin A, Wagner L, Weinberg M, Yi-Wen K, Wood E, Bradbury AR. An eHealth Delivery Alternative for Cancer Genetic Testing for Hereditary Predisposition in Patients With Metastatic Cancers: Protocol for a Randomized Trial. JMIR Res Protoc. 2025 Aug 25;14:e72515. doi: 10.2196/72515. PMID 40853717